CLINICAL TRIAL: NCT05453253
Title: Immune Response to a Delayed Second Dose of Oral Cholera Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Epicentre (Other)
Collaborators: Ministry of Health, Guinea (Other Government); Massachusetts General Hospital (Other); Médecins Sans Frontières, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OCV_DelayedProtocol
Record Dates: First submitted 2022-06-01; First posted 2022-07-12 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Cholera; Vibrio Cholerae Infection
Keywords: Delayed vaccine; Cholera; non-inferiority
MeSH Terms: conditions — Cholera | interventions — Cholera Vaccines

STUDY DESIGN:
Intervention Model Description: Considering 20% loss of follow-up and sampling failures at 14 days post 2nd OCV, the aim is to enroll 152 participants per arm for the analysis. Thus 456 (3*152) participants will be recruited. Also, participants with a blood sampling failure at baseline (pre-1st OCV) will be replaced and withdrawn before randomization. Thus 456 (3*152) participants with an appropriate blood sample at baseline will be randomisedecruited.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- interventional 6 months interval between OCV doses (Experimental): This intervention arm will modify the recommended interval for administration of the second Euvichol-Plus®, which will be extended to 6 months.
  Interventions: Biological: Delayed second dose of oral cholera vaccine, Euvichol-Plus
- interventional 12 months interval between OCV doses (Experimental): This intervention arm will modify the recommended interval for administration of the second Euvichol-Plus®, which will be extended to 12 months.
  Interventions: Biological: Delayed second dose of oral cholera vaccine, Euvichol-Plus
- control arm (standard 14-day interval) (Active Comparator): Participants will receive the oral cholera vaccine, Euvichol-Plus®, according to the manufacturer instructions: 2 doses two weeks apart.
  Interventions: Biological: Oral cholera vaccine, Euvichol-Plus, according to manufacturer notice

INTERVENTIONS:
Biological: Delayed second dose of oral cholera vaccine, Euvichol-Plus — The intervention arms (6 and 12 months) will modify the recommended interval for administration of the second vaccine dose, which will be extended to 6 and 12 months according to the intervention arm.
  Arms: interventional 12 months interval between OCV doses; interventional 6 months interval between OCV doses
Biological: Oral cholera vaccine, Euvichol-Plus, according to manufacturer notice — Euvichol-Plus, a WHO prequalified oral cholera vaccine, contains modified killed whole cell vaccine of formalin killed Vibrio cholerae strains of O1 Inaba, O1 Ogawa and O139.
  In the control arm, participants will receive the Euvichol-Plus following the manufacturer recommendations: two doses administered orally 14 days apart for individuals aged ≥1 year.
  Arms: control arm (standard 14-day interval)

SUMMARY:
Immune response to a delayed second dose of oral cholera vaccine

A randomized, controlled, non-inferiority immunogenicity trial in Conakry, The Republic of Guinea

DETAILED DESCRIPTION:
Manufacturers of oral cholera vaccine (OCV) recommend a 7- or 14-days interval between two doses. To carry out two rounds of mass vaccination within this delay is not always feasible and many campaigns implemented to date have used a longer interval. Recent evidence indicates that an extended interval between OCV doses might result in equivalent seroconversion rates and in an improved boosting of mucosal immune responses following the second dose. To guide future OCV vaccination campaigns and improve cholera prevention, it is important to demonstrate the non-inferior immune response of an extended interval between OCV doses.

The Investigators aim to demonstrate the non-inferiority of the humoral immune response between individuals receiving a second Euvichol-Plus® pre-qualified OCV dose either 6 or 12 months after the initial dose and individuals receiving a second pre-qualified OCV dose 14 days after the initial dose. The humoral immune response will be assessed as the post-vaccination titer of serum vibriocidal antibodies at 14 days post-2nd dose vaccination. Secondary outcomes include the comparison of the overall rate of vibriocidal seroconversion 14 days after either the first or the second vaccine dose. A subsample of individuals ≥ 18 years will have additional serological evaluation to characterize the kinetics of their antibody responses up to 6 months after the second OCV vaccine dose. Although the vaccine has an established and safe profile, occurrence of adverse events and serious adverse events following vaccination will be assessed (safety evaluation).

The study will be an open-label, randomized, controlled, non-inferiority immunogenicity trial comparing the humoral immune responses to OCV in two interventions arms (6 and 12 months interval between OCV doses) compared with a control arm (standard 14-day interval). In each arm, the aim is to recruit 152 individuals aged 1 to 40 year-old eligible for OCV vaccination from the general population (ie. 456 individuals in total). The sub-sample allowing characterizing the kinetics of the humoral response up to 6 months after the administration of the second dose will include 38 participants in each intervention and control arm, among the participants aged ≥ 18 years. In total, 456 individuals will be recruited.

The study will be conducted in Conakry, in the Republic of Guinea. Participants will be primarily enrolled in the commune of Dixinn on a voluntary basis. All participants in the intervention and control arms will be invited to a first visit for assessment of eligibility and 1st OCV dose, followed by a visit 14 days after the 1st OCV dose for blood sampling. According to the study arm, the 2nd OCV dose will be administered at 14 days, 6 months or 1 year after the 1st dose and will be followed by a visit 14 days later for blood sampling. Participants in the sub-study will be invited to additional study visits (up to twelve visits in total) for blood sampling. At each visit, blood will be drawn for immunologic analyses.

ELIGIBILITY:
Inclusion Criteria:

* Any healthy individual ≥ 1 year-old and younger than 40 years old , eligible for OCV vaccination (not suffering from a medical condition that contraindicates vaccination, i.e. any acute illness, including acute gastrointestinal illness or acute febrile illness).
* Living in the study area with no plan to move away over the study period (up to 18 months).
* Who provided written informed consent or whose representative (mother, father or main caretaker) provided written informed consent in case of individuals younger than 18 years. A written assent will also be obtained from adolescents (10-17 years)
* An individual who (or whose mother, father or main caretaker) is, based on the judgment of the investigator, capable of complying with the study requirements.

Exclusion Criteria:

* Known history of hypersensitivity reactions to other vaccines.
* Individual acutely ill or with signs of infection at the time of enrolment (e.g. fever > 38⁰C)
* Gastrointestinal symptoms including nausea, vomiting, diarrhea, or decreased appetite within 24 hours prior to study initiation .
* Diarrhea, administration of antidiarrheal drugs or antibiotics to treat diarrhea or abdominal pain either lasting 2 weeks or longer within 6 months prior to study initiation, or occurring during the week before study initiation.
* Other vaccination within 1 week prior to study initiation or planned vaccination during the following month after vaccine intake .
* Participation in another trial with investigational product within 1 month prior to study initiation.
* Pregnant (as determined by a urine test on the day of each vaccination) or lactating women, women of reproductive age planning pregnancy before the end of the study period (up to minimum 18 months).
* An individual thought to have difficulty participating in the study due to other reasons (such as mental disorders, alcohol or drug intoxication), based on the judgment of the investigator.
* History of cholera vaccination or history of cholera as diagnosed by a medical person in a health facility (with or without laboratory confirmation).
* Severe chronic diseases or medical conditions, based on the medical judgment of the investigator, such as known low hemoglobin level or symptomatic anemia, severe acute malnutrition, chronic infection (e.g. tuberculosis), sequel of poliomyelitis, immunodeficiency due to symptomatic HIV/AIDS.
* Based on participant verbal reporting of the participant at inclusion, more than two persons in households <5 persons or three participants in households ≥ 5 persons.
* Thrombocytopenia or bleeding disorders or other known contraindication to venipuncture. Severe medical condition that contraindicates vaccination. In particular, a) known history of immune function disorders; or b) current use of steroids cytotoxic drugs, immunosuppressant, immune modifying drug, Prednisolone, Azathioprine, Cyclosporin, Interferon, G-CSF, Tacrolimus, Everolimus, Sirolimus; or c) known active malignancy with the exception of adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years; or d) known uncompensated NYHA Class 3 or 4 congestive heart failure; or e) known myocardial infarction within the previous 6 months; or f) known neurological and/or psychiatric disorder.

Ages: 1 Year to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 456 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Serum vibriocidal antibody specific to V. cholerae O1, Inaba, Ogawa and O139 strains | 14 days after the administration of the second vaccine dose
  Serum vibriocidal antibody Geometric Mean Titre (GMT)

SECONDARY OUTCOMES:
Serum vibriocidal antibody specific to V. cholerae O1, Inaba, Ogawa and O139 strains | Just before and 14 days after administration of the first dose and and just before the second OCV dose
  Serum vibriocidal antibody Geometric Mean Titre (GMT)
Serum vibriocidal anti-OSP IgA, IgG, IgM | Just before and 14 days after administration of the first and the second OCV dose
  Serum vibriocidal anti-OSP IgA, IgG, IgM titres measured using Enzyme-linked immunosorbend essay (ELISA)
Anti-CtxB immunoglobulines | Just before and 14 days after administration of the first and the second OCV dose
  Anti-CtxB immunoglobulines titres measured using Enzyme-linked immunosorbend essay (ELISA)
Immediate Adverse Events (IAEs) (Safety) | Up to 30 minutes after each OCV dose
  All participants will be observed by clinicians for 30 minutes after each vaccination to monitor for any immediate adverse events (IAEs)
Adverse events (AEs) (Safety) | Until 14 days after the administration of the first and the second OCV dose
  Solicited and unsolicited AEs will be actively monitored by clinicians at the study visits for 14 days following administration of each vaccine dose.
Serious Adverse Events (SAEs) (Safety) | Up to end of the participants' follow-up i.e. 18months
  SAEs will be monitored by clinicians up to end of the participants' follow-up.

OTHER OUTCOMES:
Serum vibriocidal antibody specific to V. cholerae O1, Inaba, Ogawa and O139 strains | In a subgroup of participants: At 4, 7, 28 and 180 days after administration of the first and the second OCV dose
  Serum vibriocidal antibody Geometric Mean Titre (GMT)
Serum vibriocidal anti-OSP IgA, IgG, IgM | In a subgroup of participants: At 4, 7, 28 and 180 days after administration of the first and the second OCV dose
  Serum vibriocidal anti-OSP IgA, IgG, IgM titres measured using Enzyme-linked immunosorbend essay (ELISA)
Anti-CtxB immunoglobulines | In a subgroup of participants: At 4, 7, 28 and 180 days after administration of the first and the second OCV dose
  Anti-CtxB immunoglobulines titres measured using Enzyme-linked immunosorbend essay (ELISA)

CONTACTS AND LOCATIONS:
Locations (1):
- Dixinn, Conakry, Guinea